CLINICAL TRIAL: NCT06091930
Title: Phase I, Non-randomised, Open-label, Multi-centre Dose Escalation and Expansion Trial of BI 765049 and BI 765049 + Ezabenlimab Administered by Repeated Intravenous Infusion in Asian Patients With Malignant Solid Tumours Expressing B7-H6
Brief Title: A Study to Test Different Doses of BI 765049 Alone and in Combination With Ezabenlimab in Asian People With Advanced Cancer (Solid Tumours) Positive for B7-H6
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1454-0004
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Cancer; Lung Cancer; Pancreatic Cancer; Colorectal Cancer; Head and Neck Cancer; Liver Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial is divided in four parts. Part I and Part III will have a sequential assignment while Part II and Part IV will have a parallel assignment.
Masking Description: All trial parts will be conducted open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part I: BI 765049 (Experimental): BI 765049 monotherapy - dose escalation
  Interventions: Drug: BI 765049
- Part II: BI 765049 (Experimental): BI 765049 monotherapy - dose expansion
  Interventions: Drug: BI 765049
- Part III: BI 765049 + ezabenlimab (Experimental): BI 765049 + ezabenlimab combination therapy - dose escalation
  Interventions: Drug: BI 765049; Drug: Ezabenlimab
- Part IV: BI 765049 + ezabenlimab (Experimental): BI 765049 + ezabenlimab combination therapy - dose expansion
  Interventions: Drug: BI 765049; Drug: Ezabenlimab

INTERVENTIONS:
Drug: BI 765049 — BI 765049
Drug: Ezabenlimab — Ezabenlimab
  Other Names: BI 754091
  Arms: Part III: BI 765049 + ezabenlimab; Part IV: BI 765049 + ezabenlimab

SUMMARY:
This is a study in adults from Asia with different types of advanced cancer (solid tumours). People can join the study if they have cancer of the stomach, large bowel and rectum, pancreas, liver, head and neck or non-small cell lung cancer. This is a study for people for whom previous treatment was not successful or no treatment exists. People can participate if their tumour has the B7-H6 marker.

The purpose of this study is to find the highest dose of BI 765049 that people with advanced cancer can tolerate when taken (alone and) together with ezabenlimab. Another purpose is to check whether BI 765049 taken (alone and) together with ezabenlimab can make tumours shrink. Both medicines may help the immune system fight cancer.

Participants can stay in the study up to 3 years, as long as they can tolerate it and can benefit from it. During this time, they visit the study site about every 3 weeks. At the study site they get BI 765049 alone or in combination with ezabenlimab as an infusion into a vein. BI 765049 is given in 3-week cycles, ezabenlimab is given once every 3 weeks.

The doctors check the health of the participants and note any health problems that could have been caused by BI 765049 or ezabenlimab. Doctors regularly check the size of the tumour and check whether it has spread to other parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated, written inform consent form (ICF) (ICF1 for B7-H6 testing for all patients except those with colorectal cancer (CRC); ICF2 for all patients) describing the study in accordance with International Council on Harmonisation Good Clinical Practice (ICH-GCP) and local legislation prior to any trial-specific procedures, sampling, or analyses.
* ≥18 years of age at the time of signature on the ICFs (ICF1 and ICF2).
* Histologically or cytologically confirmed diagnosis of an advanced, unresectable, and/or metastatic gastrointestinal cancer, colorectal cancer, pancreatic cancer, liver cancer, head and neck cancer, or lung cancer.
* Disease progression despite conventional treatment, intolerant to or not a candidate for conventional treatment, or with a tumour for which no conventional treatment exists.
* Agree to the collection of tumour samples (as slides from archival diagnostic samples or fresh tumour biopsies) for confirmation of B7-H6 expression at Screening Visit 02 for colorectal cancer (CRC) patients or at Screening Visit 01 for all other patients.
* Confirmed B7-H6 expression on tumour tissue sample (archived or fresh tumour biopsy) based on central pathology review except for patients diagnosed with advanced or metastatic colorectal cancer (CRC).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* At least one evaluable target lesion as defined per response evaluation criteria in solid tumors (RECIST v1.1), outside of the central nervous system (CNS), separate from any lesion(s) identified for tumour biopsy. Tumour lesions that have been irradiated ≥28 days before the start of treatment, and have subsequently had documented progression, may be chosen as target lesions only in the absence of measurable lesions that have not been irradiated.
* Further inclusion criteria apply

Exclusion Criteria:

* History of a major surgery within 28 days prior to first dose of BI 765049 (major according to the Investigator's assessment).
* Previous or concomitant malignancies other than the one treated in this trial within the last 3 years except:

  * Effectively treated non-melanoma skin cancers
  * Effectively treated carcinoma in situ of the cervix
  * Effectively treated ductal carcinoma in situ
  * Other effectively treated malignancy that is considered cured by local treatment
* Known leptomeningeal disease or spinal cord compression due to disease.
* Require anticoagulant treatment which cannot be safely interrupted, if medically needed for a study procedure (e.g., biopsy) based on the opinion of the Investigator.
* Hepatitis C virus (HCV) infection, defined as:

  * Currently receiving curative antiviral treatment for HCV infection, and/or
  * HCV viral load is above the limit of quantification (HCV Ribonucleic acid (RNA) positive)
* Hepatitis B virus (HBV) infection with the following laboratory evidence: positive results of hepatitis B surface (HBs) antigen and presence of Hepatitis B core (HBc) antibody together with HBV-deoxyribonucleic acid (DNA).
* Presence of any infection requiring systemic antimicrobial treatment within 7 days prior to first dose of trial medication. Patients who have any clinical signs of infection (e.g. fever or leukocytosis) within 48 hours prior to first dose of trial medication are not eligible.
* Patients with known history of human immunodeficiency virus (HIV) infection who meet one or more of the following criteria:

  * Cluster of differentiation 4 (CD4+) count <350 cells/μL (local lab assessment)
  * Viral load >400 copies/mL (local lab assessment)
  * Not receiving antiretroviral therapy
  * Receiving established antiretroviral therapy for less than four weeks prior to the start of study treatment
  * History of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within 12 months prior to start of study treatment Patients with a history of HIV who do not meet any of the criteria above are eligible to participate, but the patient must be under the care of a HIV/Infectious Diseases specialist, or a HIV/Infectious Diseases specialist must be consulted prior to inclusion.
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2028-06-09 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
Part I: Occurrence of dose-limiting toxicity (DLTs) during the maximum tolerated dose (MTD) evaluation period for BI 765049 monotherapy | One treatment cycle, defined as 3 weeks after first administration of BI 765049 or 1 week after the administration of first full dose of BI 765049, whichever is longer
Part II: Objective response based on the response evaluation criteria in solid tumors (RECIST v1.1) | Up to month 36
  Objective response will be determined by the Investigator in patients with measurable disease and will be defined as the best overall response of complete response (CR) or partial response (PR), from the first administration of trial medication until the earliest of progressive disease (PD), death, last evaluable tumour assessment before the start of subsequent anti-cancer therapy, lost to follow-up, or withdrawal of consent.
Part III: Occurrence of dose-limiting toxicity (DLTs) during the maximum tolerated dose (MTD) evaluation period for BI 765049 in combination with ezabenlimab | From first BI 765049 administration to 1 week after the first ezabenlimab dose
Part IV: Objective response based on the response evaluation criteria in solid tumors (RECIST v1.1) | Up to month 36

SECONDARY OUTCOMES:
Part I: Maximum measured concentration of BI 765049 (Cmax) after first administration | Up to 1 day
Part I: Maximum measured concentration of BI 765049 (Cmax) after multiple administrations | Up to month 37
Part III: Maximum measured concentration of BI 765049 (Cmax) after the first administration | Up to 1 day
Part III: Maximum measured concentration of BI 765049 (Cmax) after multiple administrations | Up to month 37
Part I: Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) after the first administration | Up to 1 day
Part I: Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) after multiple administrations | Up to month 37
Part III: Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) after the first administration | Up to 1 day
Part III: Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) after multiple administrations | Up to month 37
Part I: Objective response based on the response evaluation criteria in solid tumors (RECIST v1.1) | Up to month 36
  Objective response will be determined by the Investigator in patients with measurable disease who have been treated with either BI 765049 monotherapy or BI 765049 in combination with ezabenlimab and will be defined as the best overall response of complete response (CR) or partial response (PR), according to response evaluation criteria in solid tumors (RECIST v1.1). from the first administration of trial medication until the earliest of progressive disease (PD), death, or last evaluable tumour assessment before the start of subsequent anti-cancer therapy, lost to follow-up, or withdrawal of consent.
Part III: Objective response based on the response evaluation criteria in solid tumors (RECIST v1.1) | Up to month 36
Part II: Progression free survival (PFS) | Up to month 36
  Progression free survival (PFS) will be defined as the time from first treatment administration until tumour progression according to response evaluation criteria in solid tumors (RECIST v1.1) as determined by the Investigator or death from any cause, whichever occurs earlier.
Part IV: Progression free survival (PFS) | Up to month 36
Part II: Duration of response | Up to month 36
  Duration of response will be defined as the time from a patient's first documented complete response (CR) or partial response (PR), according to response evaluation criteria in solid tumors (RECIST v1.1), until the earliest of disease progression, or death.
Part IV: Duration of response | Up to month 36
Part II: Disease control | Up to month 36
  Disease control will be defined as best overall response of complete response (CR), partial response (PR) or stable disease (SD) where best overall response is as determined by the Investigator according to response evaluation criteria in solid tumors (RECIST v1.1) from the first administration of trial medication until the earliest of progression disease (PD), death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, lost to follow-up, or withdrawal of consent.
Part IV: Disease control | Up to month 36
Part II: Objective response based on the immune response evaluation criteria in solid tumors (iRECIST) | Up to month 36
  Objective response based on immune response evaluation criteria in solid tumors (iRECIST) criteria will be determined by the Investigator in patients with measurable disease and will be defined as the best overall response of complete response (CR) or partial response (PR), from the first administration of trial medication until the earliest of immune confirmed progressive disease (PD), death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, lost to follow-up, or withdrawal of consent.
Part IV: Objective response based on the immune response evaluation criteria in solid tumors (iRECIST) | Up to month 36
Part II: Maximum measured concentration of BI 765049 (Cmax) after first administration | Up to 1 day
Part II: Maximum measured concentration of BI 765049 (Cmax) after multiple administrations | Up to month 37
Part IV: Maximum measured concentration of BI 765049 (Cmax) after first administration | Up to 1 day
Part IV: Maximum measured concentration of BI 765049 (Cmax) after multiple administrations | Up to month 37
Part II: Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) after first administration | Up to 1 day
Part II: Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) after multiple administrations | Up to month 37
Part IV: Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) after first administration | Up to 1 day
Part IV: Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) after multiple administrations | Up to month 37

CONTACTS AND LOCATIONS:
Locations (9):
- Shanghai East Hospital, Shanghai, China
- Japan (4):
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Kansai Medical University Hospital, Osaka, Hirakata
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- South Korea (2):
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com